CLINICAL TRIAL: NCT04660968
Title: Dyadic Approach To Active Living and Eating Healthy: a Randomized Controlled Trial of a Dyadic Health Behavior Change Intervention vs. Nutrition Education for Older Adult Obese Couples
Brief Title: Dyadic Approach To Active Living and Eating Healthy: The DATE Study
Acronym: DATE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Concordia University, Montreal (Other)
Collaborators: Centre de Recherche de l'Institut Universitaire de Geriatrie de Montreal (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 30011381
Record Dates: First submitted 2020-10-28; First posted 2020-12-09 (Actual); Last update posted 2023-02-22 (Actual); Status verified 2022-03

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dyadic Health Behaviour Change Intervention (Experimental): The dyadic health behaviour change intervention is a 10 sessions program provided over 16 weeks. It includes nutritional, physical activity and sedentary related information, as well as couples-based adaptation of motivational interviewing, self-monitoring, goals setting, stimulus control, problem-solving, and relapse prevention as well as specific strategies to support their partner's autonomy and intrinsic motivation.
  Interventions: Behavioral: Dyadic health behaviour change intervention
- Dyadic nutrition counselling intervention (Active Comparator): The couples-based nutrition counselling intervention is a 10 sessions program provided over 16 weeks. Topics are based on Dietitians of Canada's Practice-based Evidence in Nutrition discussions. Participants are also encouraged to meet the current physical activity recommendations. Both members of the couples are seen at the same, but no intervention target specifically the behaviour change process or the romantic relationship.
  Interventions: Behavioral: Dyadic nutrition counselling intervention

INTERVENTIONS:
Behavioral: Dyadic health behaviour change intervention — The dyadic behaviour change intervention adopts a dyadic coping perspective wherein appraisal of shared responsibility, agreement on tasks, and collaboration are fostered throughout the intervention. The intervention will target four behaviour goals: reducing overall caloric intake, substituting empty calorie foods with healthier alternatives, reducing sedentary behaviour, and increasing physical activity. The specific behavioural change strategies will include motivational interviewing, self-monitoring, goal setting, stimulus control, problem solving, and relapse prevention. Each session will also include a short education component on healthy eating to improve participants' adherence to the updated Canada's Food Guide. Participants will have access to web-based exercise training sessions. Intervention sessions will be delivered online.
  Arms: Dyadic Health Behaviour Change Intervention
Behavioral: Dyadic nutrition counselling intervention — The couples-based education nutrition intervention will provide extensive information on healthy eating. However, it will not include any behavioural change principles. Topics will be based on Dietitians of Canada's Practice-based Evidence in Nutrition (PEN) discussions in the database that focus on healthy eating for older adults. The topics covered will include increasing fruits and vegetables, hidden (empty) calories, how to read food labels, portion control, reducing salt and saturated fat, plant-based proteins, and eating for healthy bones. Participants in this group will also be told to increase their levels of physical activity to 150 minutes of moderate to vigorous physical activity per week, as per the Canadian Guidelines. Participants will have access to web-based exercise training sessions. However, physical activity will not be discussed explicitly during the intervention. Intervention sessions will be delivered online.
  Arms: Dyadic nutrition counselling intervention

SUMMARY:
The purpose of the DATE study is to evaluate the feasibility and acceptability and a preliminary evaluation of the efficacy of a dyadic health behaviour change intervention to improve healthy eating, physical activity, and dyadic coping among older obese couples. This novel intervention will use a dyadic adaptation of common health behaviour change strategies and will promote a dyadic coping approach to health behaviour change that emphasize partners' interdependence and shared responsibility for the creation of a home environment conducive to a healthy lifestyle. For this project 35 obese older adults cohabiting dyads will be randomized to either the couples-based dyadic health behaviour change intervention or a couples-based nutrition counselling control condition.

ELIGIBILITY:
Inclusion Criteria:

* At least one of the partners is retired
* Partners cohabitating for at least 2 years.
* Obesity: BMI between 30-45 kg/m2

Exclusion Criteria:

1. Currently enrolled in a weight loss program
2. On a special diet
3. Eating disorder
4. Uncontrolled diabetes
5. Stroke
6. Heart problems (heart attack, heart failure, surgery of the heart or of the carotid arteries, pacemaker)
7. Other medical issues or medical treatment that would prevent doing physical activity

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2020-12-15 (Actual); Primary Completion 2023-06-15 (Estimated); Study Completion 2024-11-15 (Estimated)

PRIMARY OUTCOMES:
Change in Healthy Eating Index | Baseline, 4 months, 7 months, 16 months
  Canadian adaptation of the Healthy Eating Index based on a 3-day food diary

SECONDARY OUTCOMES:
Change in Moderate-to-Vigorous Physical Activity (minutes per day) | Baseline, 4 months, 7 months, 16 months
  Objective physical activity assessed using accelerometry for 7 consecutive days.
Change in self-reported physical Activity | Baseline, 4 months, 7 months, 16 months
  Self-reported physical activity assessed using the Physical Activity Scale for the Elderly (total score ranges from 0 to 793, with higher scores indicating greater physical activity).
Change in weight (kg) | Baseline, 4 months, 7 months, 16 months
  Body weight assessed using a digital scale
Change in waist circumference (cm) | Baseline, 4 months, 7 months, 16 months
  Waist circumference assessed using a measuring tape anchored at the top of the hip bone.
Change in Relationship Satisfaction | Baseline, 4 months, 7 months, 16 months
  Relationship satisfaction assessed using the Couples Satisfaction Index-4 (total score ranges from 0-21, with higher scores indicating greater relationship satisfaction).
Change in Dyadic Coping | Baseline, 4 months, 7 months, 16 months
  Dyadic coping assessed using the Common Dyadic Coping subscale of the Dyadic Coping Inventory (total score ranges from 0-30, with higher scores indicating common more dyadic coping).
Change in Spousal Social Support for Diet | Baseline, 4 months, 7 months, 16 months
  Diet social support assessed using the spousal version of the Social Support for Diet (total score ranges from 0 to 50 with higher scores indicating greater social support for diet).
Change in Spousal Social Support for Exercise | Baseline, 4 months, 7 months, 16 months
  Spousal social support for exercise assessed using the spousal version of the Social Support for Exercise scale (total score ranges from 0 to 60 with higher scores indicating greater social support for exercise).
Change in Communal Coping | Baseline, 4 months, 7 months, 16 months
  Communal coping assessed using a home-made communal coping scale (total score range from 6-60 with higher score indicating greater communal coping).
Change in Autonomy Support | Baseline, 4 months, 7 months, 16 months
  Autonomy support assessed using the spousal version for the Important Other Climate Questionnaire (total scores 6-42, with higher scores indicating more autonomy support).

OTHER OUTCOMES:
Changes in Self-Efficacy for Exercise | Baseline, 4 months, 7 months, 16 months
  Self-Efficacy for Exercise assessed using the Self-Efficacy for Exercise Scale (total score ranges from 5-25, with higher score indicating greater exercise self-efficacy).
Changes in Self-Efficacy for Diet | Baseline, 4 months, 7 months, 16 months
  Self-Efficacy for Diet assessed using the Weight Efficacy LifeStyle Questionnaire (total score ranges from 0-180, with higher score indicating greater diet self-efficacy).
Changes in Action Planning | Baseline, 4 months, 7 months, 16 months
  Action planning assessed using a home-made questionnaire based on the Health Action Process Approach (total score ranges from 0-54, with greater score indicating more action planning).
Changes in Functional Fitness | Baseline, 4 months, 7 months, 16 months
  Functional fitness assessed using the Short Physical Performance Battery (total score ranges from 0-12 with higher score indicating better functional fitness).
Changes in Maximal Handgrip Strength (kg) | Baseline, 4 months, 7 months, 16 months
  Maximal handgrip strength assessed using a hand dynamometer.
Changes in Depressive Symptoms | Baseline, 4 months, 7 months, 16 months
  Depressive symptoms assessed using the Center for Epidemiological Study-Depression (total score ranges 0 to 60, with higher score indicating more depressive symptoms)
Changes in Sleep Quality | Baseline, 4 months, 7 months, 16 months
  Sleep quality assessed using Pittsburgh Sleep Quality Index (total score ranges 0 to 21, with higher score indicating poorer sleep quality)

CONTACTS AND LOCATIONS:
Locations (1):
- Concordia University, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No
Anonymized study data available upon request